CLINICAL TRIAL: NCT03618602
Title: A Phase I Study to Evaluate the Safety, Pharmacokinetics and Efficacy of Bisthianostat in Refractory or Recurrent Multiple Myeloma Patients
Brief Title: Safety, Pharmacokinetics and Efficacy Study of Bisthianostat in Refractory or Recurrent Multiple Myeloma Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Theorion Pharmaceutical Co Ltd. (Industry)
Collaborators: Shanghai Institute of Materia Medica, Chinese Academy of Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CH-020PI
Record Dates: First submitted 2018-07-13; First posted 2018-08-07 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Refractory Multiple Myeloma; Recurrent Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 100mg Bisthianostat (Experimental): 100mg starting dose taken orally on Day 1, 4,7,11,14,18,21,25 and 28 of each cycle(4 weeks).
  Interventions: Drug: Bisthianostat
- 200mg Bisthianostat (Experimental): 200mg Bisthianostat taken orally on Day 1, 4,7,11,14,18,21,25 and 28 of each cycle(4 weeks).
  Interventions: Drug: Bisthianostat
- 400mg Bisthianostat (Experimental): 400mg Bisthianostat taken orally on Day 1, 4,7,11,14,18,21,25 and 28 of each cycle(4 weeks).
  Interventions: Drug: Bisthianostat
- 600mg Bisthianostat (Experimental): 600mg Bisthianostat taken orally on Day 1, 4,7,11,14,18,21,25 and 28 of each cycle(4 weeks).
  Interventions: Drug: Bisthianostat

INTERVENTIONS:
Drug: Bisthianostat — Bisthianostat is a histone deacetylase inhibitor (HDAC inhibitor) for the treatment of multiple myeloma.
  Other Names: CF367-C, CFH367-C, CF367, PY-1

SUMMARY:
This is a first-in-human study to investigate the safety, tolerability, pharmacokinetics, and efficacy of Bisthianostat in refractory or recurrent multiple myeloma patients.

DETAILED DESCRIPTION:
This is a first-in-human, single center, open-label, single arm, dose escalating phase I study. This study will be conducted in 3 parts.

Phase A : Patients will receive single dose of bisthianostat to evaluate the single-dose pharmacokinetics and safety.

Phase B: After single-dose phase, patients will receive multiple dose bisthianostat for 4 weeks on day 1,4,11,14,18,21,25,28 to evaluate the multiple-dose pharmacokinetics and safety

Phase C: Patients will continue on the study if they benefit from the drug and not experience any serious side effects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as stage II or III (Durie-Salmon Staging System) multiple myeloma with disease progression or recurrence after at least two cycles of systemic antimyeloma treatment.
* Serum M protein≥ 5.0g / L, or urine M protein ≥ 200mg / 24h, or serum free light chain ≥ 200mg / L.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2.
* Expected survival of ≥3 months.
* Female participants of childbearing potential should have negative urine pregnancy test in screening period (accept previous test result within 14 days before screening), and must agree to adopt effective contraceptive measures within 14 days before receiving first dose of study drug, during the treatment period and within 28 days after final dose of study drug.
* Male participants must agree to adopt effective contraceptive measures and not allowed to donate sperms during the treatment period, and within 28 days after final dose of study drug.
* Hemoglobin ≥ 80 g/L, Platelet≥50×109/L (50,000/mm3), Absolute Neutrophil Count≧1.0×109/L (1000 cells/mm3), Prothrombin time(PT) and activated partial thromboplastin time ≤ 2 x Upper Limit of Normal (ULN)
* AST or ALT ≤ 1.5 x ULN, total bilirubin≤ 1.5 x ULN;
* Serum Creatinine ≤ 1.5 x ULN, glomerular filtration rate≥ 50 ml/min;
* NYHA Class I or II
* Written informed consent obtained prior to participation in the study

Exclusion Criteria:

* Pregnant or lactating women.
* Non-secretory multiple myeloma patients.
* Plasma cell leukemia patients.
* Received any anti-cancer medication or experimental drugs against multiple myeloma within 1 week before first dose of bisthianostat, any experimental treatment other than medication (eg. leukocyte donor/monocyte infusion) within 56 days before first dose of bisthianostat. Participation in any other drug or medical devices within 56 days before the study.
* Stem cell transplant planned on the following 28 days.
* Uncontrolled hypercalcemia after treatments, eg. saline infusion.
* Renal insufficiency required hemodialysis or peritoneal dialysis.
* NCI-CTCAE grade 2 Peripheral Neuropathy.
* Serious heart disease in the past 6 months, including angina requiring surgery, uncontrolled hypertension after anti-hypertensive treatments (Systolic blood pressure> 160 mmHg, Diastolic blood pressure>90mmHg); Myocardial infarction; Grade II-IV congestive heart failure; unstable angina.
* HIV, HCV or HBV (HBV-DNA > 20 IU/mL) infection.
* Patients with any other prior malignancy, except for skin basal cell carcinoma, cervical carcinoma in situ, breast carcinoma in situ, skin squamous cell carcinoma that have been treated and controlled.
* Imaging evidences show tumors have involved main blood vessels and nerves.
* Patients with significant central nervous system lesions.
* Patients with mental illness.
* Patients with history of alcohol or drug abuse, patients with allergy to the active ingredient or excipients of study drug, and patients who are unable or unwilling to receive the intravenous administration.
* Active infection (Bacteria, fungi, virus etc), fever with body temperature > 38 ℃ for reasons unknown.
* Other situations that investigator considers it's inappropriate for patients to participate in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-04-25 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose of Bisthianostat | Up to 24 months
  To determine the maximum tolerated dose of Bisthianostat in refractory or recurrent multiple myeloma patients.
Treatment-related adverse events considered as dose-limiting toxicity | During the first cycle (4 weeks)
  To evaluate the severity of treatment-related AEs considered as dose-limiting toxicity.

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) | During the first cycle (4 weeks)
  To determine the Peak Plasma Concentration of Bisthianostat.
Area under the plasma concentration versus time curve (AUC) | During the first cycle (4 weeks)
  To determine the Area under the plasma concentration versus time curve of Bisthianostat.
Time of Peak Concentration (Tmax) | During the first cycle (4 weeks)
  To determine the time of peak concentration of Bisthianostat.
Half life (T1/2) | During the first cycle (4 weeks)
  To determine the half-life of Bisthianostat.
Objective Response Rate | Up to 1 month after last dose
  To evaluate the objective response rate in refractory or recurrent myeloma patients after bisthianostat treatments.
Incidence of adverse events related to treatments | Up to 1 month after last dose
  To evaluate the incidence of adverse events that are related to treatments in refractory or recurrent myeloma patients
Incidence of laboratory abnormalities related to treatments | Up to 1 month after last dose
  To evaluate the incidence of laboratory abnormalities that are related to treatments in refractory or recurrent myeloma patients

CONTACTS AND LOCATIONS:
Overall Officials: Jian Hou, MD, Principal Investigator — RenJi Hospital
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China